CLINICAL TRIAL: NCT03086109
Title: The Prevalence of Bone Degenerative Diseases in Beijing - a Cross-sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Wei Tian, President, Beijing Jishuitan Hospital
Other Study IDs: 2012BAI10B02-Cohort
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Cross-sectional Study; Degenerative Disease Joint; Degenerative Disc Disease
Keywords: prevalence; Bone Degenerative Disease
MeSH Terms: conditions — Joint Diseases; Intervertebral Disc Degeneration | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Risk factors — Risk factors associated bone degenerative diseases

SUMMARY:
The purpose of this observational study is to investigate the prevalence and risk factors of bone degenerative diseases

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years， residents of Beijing city
2. Must demonstrate willingness to participate in the study by signing the written informed consent

Exclusion Criteria:

1. Subjects who had surgery on disc or knee
2. Pregnent women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The residents of Beijing voluntary to participant to this study
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of bone degenerative diseases | 1 year
  Degree of disc and knee degeneration based on imaging examination (etc. CT OR MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tian, MD, Study Director — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, China